CLINICAL TRIAL: NCT01781156
Title: Effect of Reducing Phosphorus Absorption on Cardiac Biomarkers in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ai Peng, Director of the department of Nephrology, Shanghai 10th poeple's hospital, Shanghai 10th People's Hospital
Other Study IDs: 2012RES-047; 81270136 (Other Grant/Funding Number: China NNSF)
Record Dates: First submitted 2013-01-24; First posted 2013-01-31 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2014-11

CONDITIONS: End Stage Renal Failure
Keywords: phosphorus; hemodialysis; cardiac biomarkers
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hyperphosphatemia and elevated cardiac biomarkers are two key characteristics of patients in end stage renal diseases(ESRD),however the majority of whom are in the absence of acute coronary syndrome(ACS). And it is still unclear why cardiac biomarkers would increase in those patients. We hypothesized that excessive phosphorus is account for that phenomenon.To confirm that hypothesis,we used one phosphorus binder to reduce phosphorus absorption in hemodialysis patients for some time and observed the change of cardiac biomarkers of those patients.

DETAILED DESCRIPTION:
Cardiovascular disease is one of the leading causes of morbidity and mortality in patient with chronic kidney disease(CKD), accounting for more than 50% of all deaths.When myocardial cells get injured, cardiac biomarkers will be released into the circulation. Elevated cardiac biomarkers have been observed in patients with various degrees of renal failure. However, the majority of those CKD patients are in the absence of acute coronary syndrome. So far, it is still unclear the mechanisms of the increased biomarkers in CKD patients. Meanwhile, hyperphosphatemia is one of the major features of CKD, particularly of end stage renal disease(ESRD). Lots of evidences have shown that high levels of serum phosphorus and an elevation of the serum calcium × phosphorus product can lead to cardiovascular calcifications and subsequent cardiovascular morbidity and mortality in patients with CKD.it is tempting to hypothesize that hyperphosphatemia may be responsible for the rise of cardiac biomarkers in CKD patients.So we use one phosphate binder to reduce phosphorus absorption in hemodialysis patients for one year and observe the change of cardiac biomarkers of those patients.

ELIGIBILITY:
Inclusion Criteria:

* Time of receiving hemodialysis is more than 1 year;
* Hyperphosphatemia before hemodialysis;
* Never use any phosphorus binder in the past 6 months.

Exclusion Criteria:

* Receiving coronary artery stent implantation before;
* Having any cardiovascular disease in the past 6 months;
* Cannot tolerate the side effects of phosphorus binder;
* Dose not take medicine according to the prescription;
* inadequate dialysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from patients of nephrology department of Shanghai 10th people's hospital in Shanghai,China.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2017-02 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Reducing cardiac biomarkers in hemodialysis patients | 6 months

SECONDARY OUTCOMES:
Improving cardiac function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ai Peng, Ph.D,M.D, Principal Investigator — Shanghai 10th People's Hospital of Tongji University
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, China